CLINICAL TRIAL: NCT00051948
Title: Phase 1-2a Dose-Ranging Study of TLK286 in Combination With Paraplatin (Carboplatin) in Recurrent Ovarian Cancer
Brief Title: TLK286 in Combination With Paraplatin (Carboplatin) in Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Gail Brown, M.D. Chief Medical Officer, Telik, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.2018
Record Dates: First submitted 2003-01-17; First posted 2003-01-22 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2007-02

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — TER 286

INTERVENTIONS:
Drug: TLK286

SUMMARY:
This is a dose-ranging, open label, Phase 1-2a study of TLK286 in combination with Paraplatin (carboplatin) in patients with recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed diagnosis of epithelial cancer of the ovary, fallopian tube, or primary peritoneal cancer
* Recurrent ovarian cancer or persistent disease following primary treatment
* At least one, but no more than four, prior chemotherapy regimens (all platinum-containing counted as one)
* At least 18 years of age

Exclusion Criteria

* Pregnant or lactating women
* History of prior malignancy except for adequately treated carcinoma in situ of the uterine cervix, basal cell or squamous cell skin cancer, or other cancer for which patient has been disease-free for at least 2 years
* Known leptomeningeal metastases or carcinomatous meningitis
* Having received whole pelvis radiation therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2003-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Santa Monica Hematology/Oncology Consultants, Santa Monica, California
  - Midwest Cancer Research Group, Inc., Skokie, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - M.D. Anderson Cancer Center, Houston, Texas